CLINICAL TRIAL: NCT07030712
Title: A Phase 1 Open-label Study to Evaluate the Safety and Efficacy of MK-8294 Monotherapy in Advanced Solid Tumors
Brief Title: A Clinical Study of MK-8294 in Participants With Advanced Solid Tumors (MK-8294-001)
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Merck Sharp & Dohme LLC (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: 8294-001; 2024-516870-31-00 (Registry Identifier: EU CT); U1111-1311-2807 (Registry Identifier: UTN); MK-8294-001 (Other: Merck)
Record Dates: First submitted 2025-06-12; First posted 2025-06-22 (Actual); Last update posted 2025-10-30 (Actual); Status verified 2025-10

CONDITIONS: Metastatic Neoplasm
Keywords: Metastases; Neoplasm
MeSH Terms: conditions — Neoplasm Metastasis; Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- MK-8294 (Experimental): Participants will receive MK-8294 monotherapy in escalating doses starting from 30 µg up to a planned 70 mg via intravenous (IV) infusion. In addition, intermediate doses may also be assessed. MK-8294 will be administered on Day 1, Day 8, and Day 15 of each cycle (each cycle = 21 days). Per protocol treatment of MK-8294 has no maximum number of cycles. Participants will be treated until any of the criteria for discontinuation of study intervention are met.
  Interventions: Drug: MK-8294

INTERVENTIONS:
Drug: MK-8294 — 30 µg via intravenous (IV) infusion
  Other Names: DAB014236
Drug: MK-8294 — 100 µg via intravenous (IV) infusion
  Other Names: DAB014236
Drug: MK-8294 — 300 µg via intravenous (IV) infusion
  Other Names: DAB014236
Drug: MK-8294 — 1 mg via intravenous (IV) infusion
  Other Names: DAB014236
Drug: MK-8294 — 3 mg via intravenous (IV) infusion
  Other Names: DAB014236
Drug: MK-8294 — 10 mg via intravenous (IV) infusion
  Other Names: DAB014236
Drug: MK-8294 — 30 mg via intravenous (IV) infusion
  Other Names: DAB014236
Drug: MK-8294 — 70 mg via intravenous (IV) infusion
  Other Names: DAB014236

SUMMARY:
MK-8294, the study medicine, is a type of targeted therapy designed to treat certain solid tumors. The main goals of this study are to learn about the safety of MK-8294 and if people can tolerate it and find the highest dose level of MK-8294 that people can tolerate.

ELIGIBILITY:
Inclusion Criteria:

The main inclusion criteria include but are not limited to the following:

* Has histologically or cytologically confirmed advanced/metastatic solid tumor; including head and neck squamous cell carcinoma, cervical squamous cell carcinoma, esophageal squamous cell carcinoma, breast cancer (triple negative breast cancer, Estrogen Receptor [ER]/progesterone receptor +, human epidermal growth factor receptor 2 negative [HER2-]), endometrial, and bladder cancer by pathology report and have received, or been intolerant to/failed, all treatment known to confer clinical benefit
* Human immunodeficiency virus (HIV)-infected participants must have well controlled HIV on antiretroviral therapy (ART)
* Participants who are hepatitis B surface antigen (HBsAg) positive are eligible if they have received Hepatitis B virus (HBV) antiviral therapy for at least 4 weeks, and have undetectable HBV viral load
* Participants with history of hepatitis C virus (HCV) infection are eligible if HCV viral load is undetectable

Exclusion Criteria:

The main exclusion criteria include but are not limited to the following:

* HIV-infected participants with a history of Kaposi's sarcoma and/or Multicentric Castleman's Disease
* Has a history of New Yok Heart Association Class II or greater heart failure
* Has received any prior immunotherapy and was discontinued from that treatment due to a Grade 3 or higher immune-related Adverse Event (irAE) (except endocrine disorders that can be treated with replacement therapy) or was discontinued from that treatment due to Grade 2 myocarditis or recurrent Grade 2 pneumonitis
* Has ongoing radiation-related toxicities, requiring corticosteroids
* Has known additional malignancy that is progressing or has required active treatment within the past 2 years
* Has known active central nervous system (CNS) metastases and/or carcinomatous meningitis
* Has active autoimmune disease that has required systemic treatment in the past 2 years except replacement therapy (eg, thyroxine, insulin, or physiologic corticosteroid)
* Has history of (noninfectious) pneumonitis/interstitial lung disease that required steroids or has current pneumonitis/interstitial lung disease
* Has active infection requiring systemic therapy
* Has history of stem cell/solid organ transplant
* Has not adequately recovered from major surgery or have ongoing surgical complications

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 47 (Estimated)
Dates: Start 2025-07-23 (Actual); Primary Completion 2027-08-23 (Estimated); Study Completion 2027-08-23 (Estimated)

PRIMARY OUTCOMES:
Number of participants who experience one or more dose-limiting toxicities (DLTs) | Up to approximately 35 days
  DLT is defined as any drug-related adverse event (AE) observed during the DLT evaluation period (up to 35 days) that results in a change to a given dose or a delay in initiating the next treatment and reported as the number of participants experiencing a DLT.
Number of Participants Who Experience an Adverse Event (AE) | Up to approximately 2 years
  An AE is any untoward medical occurrence in a participant, temporally associated with the use of study treatment, whether or not considered related to the study treatment. The number of participants who experience an AE will be reported.
Number of Participants Who Discontinue Study Intervention Due to an AE | Up to approximately 2 years
  An AE is any untoward medical occurrence in a participant, temporally associated with the use of study treatment, whether or not considered related to the study treatment. The number of participants who discontinue study/study treatment due to an AE will be reported.

SECONDARY OUTCOMES:
Objective Response Rate (ORR) | Up to approximately 2 years
  ORR is defined as the percentage of participants with Complete Response (CR: disappearance of all target lesions) or Partial Response (PR: at least a 30% decrease in the sum of diameters of target lesions) per Response Evaluation Criteria in Solid Tumors Version 1.1 (RECIST). The percentage of participants who experience CR or PR as assessed by the investigator will be presented.
Area Under the Plasma Concentration-Time Curve (AUC) of MK-8294 | Predose and at designated timepoints in each cycle for up to approximately 2 years (each cycle = 3 weeks)
  Blood samples collected pre-dose and at multiple timepoints post-dose will be used for the determination of Area Under the Concentration-Time Curve of MK-8294.
Minimum Concentration (Cmin) of MK-8294 | Predose and at designated timepoints in each cycle for up to approximately 2 years (each cycle = 3 weeks)
  Cmin is defined as the lowest concentration of MK-8294 after administration of MK-8294. Blood samples collected pre-dose and at multiple timepoints post-dose will be used for the determination of Cmin of MK-8294.
Maximum Plasma Concentration (Cmax) of MK-8294 | Predose and at designated timepoints in each cycle for up to approximately 2 years (each cycle = 3 weeks)
  Cmax is defined as the peak concentration of MK-8294 after administration of MK-8294. Blood samples collected pre-dose and at multiple timepoints post-dose will be used for the determination of Cmax of MK-8294.
Time to Maximum Plasma Concentration (Tmax) of MK-8294 | Predose and at designated timepoints in each cycle for up to approximately 2 years (each cycle = 3 weeks)
  Tmax is defined as the time to reach Cmax. Blood samples collected pre-dose and at multiple timepoints post-dose will be used for the determination of Tmax of MK-8294.
Incidence of Antidrug Antibodies (ADA) to MK-8294 | Predose and at designated timepoints in each cycle for up to approximately 2 years (each cycle = 3 weeks)
  Blood samples will be collected pre-dose and at designated time points to determine the ADA response to MK-8294. The incidence of ADAs over time will be presented.
Titer of ADA to MK-8294 | Predose and at designated timepoints in each cycle for up to approximately 2 years (each cycle = 3 weeks)
  Blood samples will be collected pre-dose and at designated time points to determine the ADA titers to MK-8294.

CONTACTS AND LOCATIONS:
Overall Officials: Medical Director, Study Director — Merck Sharp & Dohme LLC
Locations (5):
- Northwestern University ( Site 0101), Chicago, Illinois, United States
- Israel (2):
  - Rambam Health Care Campus ( Site 0201), Haifa
  - Sheba Medical Center ( Site 0200), Ramat Gan
- Netherlands (2):
  - Radboudumc ( Site 0301), Nijmegen, Gelderland
  - Nederlands Kanker Instituut - Antoni van Leeuwenhoek - NKI-AVL ( Site 0300), Amsterdam, North Holland

IPD SHARING:
Plan to Share IPD: Yes
https://trialstransparency.msdclinicaltrials.com/pdf/ProcedureAccessClinicalTrialData.pdf
URL: https://externaldatasharing-msd.com/

REFERENCES:
- See also: Merck Clinical Trials Information — https://www.merckclinicaltrials.com/